CLINICAL TRIAL: NCT00443755
Title: Effect of Insulin Sensitizer Therapy on Atherothrombotic and Inflammatory Profiles Associated With Insulin Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Takeda Pharmaceuticals North America, Inc. (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-004002; R01DK041973 (NIH); KL2RR024151 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2007-02-26; First posted 2007-03-06 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes; Insulin Resistance; Metabolic Syndrome
Keywords: Inflammatory cytokine; Cardiovascular Disease; Thrombotic factors; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Metabolic Syndrome; Cardiovascular Diseases; Dyslipidemias | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Sensitizer Therapy (Active Comparator): Two insulin sensitizing drugs will be taken together for 3 months; metformin 1000 mg twice daily plus pioglitazone 45 mg daily.
  Interventions: Drug: metformin; Drug: pioglitazone
- Placebo (Placebo Comparator): Placebo tablets were used to match the active comparator drugs and dosing regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: metformin — To minimize side effects the metformin will be initiated at 500 mg twice daily with meals and increased to 1 gm twice daily with meals after two weeks and continue to a total of 3 months of dosing.
  Other Names: Fortamet; Glucophage; Glucophage Extended Release (XR); Glumetza; Riomet
  Arms: Insulin Sensitizer Therapy
Drug: pioglitazone — To minimize side effects, the pioglitazone will be initiated at 30 mg daily and increased to 45 mg daily after two weeks, and continue to a total of 3 months of dosing.
  Other Names: Actos
  Arms: Insulin Sensitizer Therapy
Drug: Placebo — Placebo tablets matching the metformin and pioglitazone tablets are given in the same regimen as the active drug arm for 3 months.
  Arms: Placebo

SUMMARY:
The objective of this study is to determine whether targeted pharmacological improvement of insulin sensitivity will normalize the associated elevations of thrombotic and inflammatory cardiovascular disease (CVD) biomarkers in individuals with insulin resistance.

DETAILED DESCRIPTION:
Individuals with diabetes mellitus (DM) are disproportionately affected by atherothrombotic disorders, including cardiovascular, cerebrovascular, and peripheral vascular diseases. Atherothrombotic disease risk and mortality are also increased with metabolic syndrome, a constellation of risk factors present in more than 34% of adults, even in absence of diabetes. Yet, large clinical trials of diabetes therapies have shown that conventional cardiovascular disease (CVD) risk factors, specifically hyperglycemia and hypertension, do not fully account for increased CVD risk associated with DM.

There may be an etiologic link among insulin resistance, inflammation and thrombotic events. This study seeks to determine if certain two diabetes medications (the insulin sensitizing medications) will affect certain biomarkers (or laboratory tests) for CVD in individuals with untreated DM or impaired fasting glucose.

Patients will be screened for inclusion into this this double-blinded, randomized), placebo-controlled study. If inclusion criteria are met and exclusion criteria not met, patients will be enrolled in the the study. Half of the subjects will be randomized (like the flip of a coin) to take two insulin sensitizing, anti-diabetic drugs pioglitazone (Actos) and metformin (Glucophage) taken together for three months and the other half of the subjects will take corresponding placebo (dummy) tablets.

Laboratory measurements will be obtained on the morning(s) following the two in-patient overnight stays in the Mayo Clinic Clinical Research Unit. The first stay will be at baseline and the second stay will be 3 months after baseline. Insulin sensitivity will be measured in the morning following a standardized meal the preceding night, and after an overnight fast.

The changes (from baseline to 3 months) in insulin sensitivity, glycemic control, the lipid profile, thrombotic markers and inflammatory markers will be determined and compared between the two arms of the study (placebo versus insulin sensitizing drugs).

ELIGIBILITY:
Inclusion criteria:

* We will study 30 patients with Type 2 Diabetes or impaired fasting glucose (15 men & 15 women) who are > 20 years old.
* Only patients who use lifestyle modification to manage their diabetes and are not on any oral hypoglycemic agents or insulin will be included.
* We will enroll subjects who have fasting glucose concentration greater than 100 mg/dl on two consecutive occasions and have a Body Mass Index between 27-36 kg/m^2.

Exclusion Criteria:

* We will exclude patients whose blood glucose is above 180 mg/dl. This will avoid the need to perform home glucose monitoring and the potential of unblinding the study by the volunteers.
* Patients taking oral hypoglycemic agents or insulin would be excluded.
* Any diseases such as active cardiovascular disease, liver diseases, kidney failure (males with serum creatinine >= 1.5mg/dl, females >=1.4 mg/dl), active endocrinopathies, debilitating chronic disease, anemia, symptoms of undiagnosed illness, history of alcoholism (alcohol use > 4oz/day) or substance abuse, chronic neurological diseases including Alzheimer's disease, stroke, etc, myopathies or any other active disease that may potentially affect the outcome measures.
* Patients on medicines such as beta blockers, corticosteroids, tricyclics, benzodiazepines, opiates, barbiturates, anticoagulants and any other drugs or preparations that may affect mitochondrial function will be excluded.
* People allergic to any of the class of drug such as lidocaine will also be excluded.
* People with pacemakers, certain aneurysm clips and claustrophobia will also be excluded as they cannot undergo magnetic resonance imaging.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] McCoy RG, Irving BA, Soop M, Srinivasan M, Tatpati L, Chow L, Weymiller AJ, Carter RE, Nair KS. Effect of insulin sensitizer therapy on atherothrombotic and inflammatory profiles associated with insulin resistance. Mayo Clin Proc. 2012 Jun;87(6):561-70. doi: 10.1016/j.mayocp.2012.02.014. PMID 22677076
- [Derived] Irving BA, Carter RE, Soop M, Weymiller A, Syed H, Karakelides H, Bhagra S, Short KR, Tatpati L, Barazzoni R, Nair KS. Effect of insulin sensitizer therapy on amino acids and their metabolites. Metabolism. 2015 Jun;64(6):720-8. doi: 10.1016/j.metabol.2015.01.008. Epub 2015 Jan 22. PMID 25733201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 8/19/2005 and 8/24/2010 at the Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 48 Northern European Americans were assessed for eligibility and of those, 20 did not meet inclusion criteria.
Groups:
- Insulin Sensitizer Therapy: Two insulin sensitizing drugs will be taken together for 3 months; metformin 1000 mg twice daily plus pioglitazone 45 mg daily. The number of subjects analyzed for baseline measures and outcome measures were the 12 subjects who completed the study.
- Placebo: Placebo tablets were used to match the active comparator drugs and dosing regimen. The number of subjects analyzed for baseline measures and outcome measures were the 13 subjects who completed the study.
Period: Overall Study
Arm/Group | Insulin Sensitizer Therapy | Placebo
Started | 14 | 14
Completed | 12 | 13
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are reported for the subjects who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Sensitizer Therapy | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 52.5 (15.6) | 52.2 (18.2) | 52.4 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25
Body Mass Index [Mean (Standard Deviation); unit: kilograms/m^2] — Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared.
  kilograms/m^2 | 32.43 (5.65) | 29.67 (3.34) | 31.00 (4.71)
Fat-Free Mass [Mean (Standard Deviation); unit: Kilograms] | 48.81 (14.29) | 46.67 (13.54) | 47.70 (13.66)
Body Fat [Mean (Standard Deviation); unit: Percentage of body weight] | 46.49 (5.92) | 43.26 (9.17) | 44.81 (7.80)
Fasting Blood Glucose [Mean (Standard Deviation); unit: milligrams per deciliter] | 126.25 (21.87) | 129.00 (26.32) | 127.68 (23.82)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage] — The HbA1c level reflects the average glucose (blood sugar) concentration over the previous 3 month period.
  Percentage | 5.97 (0.71) | 6.25 (0.65) | 6.11 (0.68)
Glucose Infusion Rate (GIR) [Mean (Standard Deviation); unit: micromols/kilogram of FFM/minute] — FFM is Fat Free Mass
  micromols/kilogram of FFM/minute | 22.28 (14.67) | 23.40 (15.27) | 22.86 (14.68)
Insulin level [Mean (Standard Deviation); unit: micro International Units per milliliter] | 15.68 (9.75) | 10.18 (5.70) | 12.82 (8.23)
Lipid Profile [Mean (Standard Deviation); unit: milligrams per deciliter]
  Triglycerides | 131.42 (54.76) | 135.00 (51.36) | 133.28 (51.93)
  High Density Lipoprotein-Cholesterol (HDL-C) | 43.33 (12.78) | 39.23 (8.74) | 41.20 (10.84)
  Non-HDL-Cholesterol | 135.58 (26.17) | 132.46 (21.65) | 133.96 (23.47)
Fibrinogen [Mean (Standard Deviation); unit: milligrams per deciliter] | 393.67 (78.63) | 418.92 (100.23) | 406.80 (89.57)
Plasminogen Activator Inhibitor 1 (PAI-1) [Mean (Standard Deviation); unit: nanograms per milliliter] | 81.83 (22.01) | 55.85 (33.70) | 68.3 (31.1)
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: milligrams per deciliter] | 0.42 (0.43) | 0.43 (0.49) | 0.42 (0.45)
Interleukin-6 (IL-6) [Mean (Standard Deviation); unit: picograms per milliliter] | 2.46 (1.68) | 3.28 (4.79) | 2.88 (3.59)
Tumor Necrosis Factor-alpha (TNF-α) [Mean (Standard Deviation); unit: picograms per milliliter] | 1.39 (0.57) | 2.98 (5.39) | 2.22 (3.91)
Adiponectin [Mean (Standard Deviation); unit: milligrams per milliliter] | 6.08 (2.17) | 5.22 (2.13) | 5.63 (2.15)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Sensitivity as Measured by Glucose Infusion Rate (GIR)
Description: Insulin sensitivity was measured the morning after an overnight fast during an in-patient stay in the Clinical Research Unit & was determined by the mean GIR necessary to maintain euglycemia during a hyperinsulinemic (1.5 mcIU/kg of FFM per minute)-euglycemic (85-95 mg/dL) clamp. The clamp is an 8 hour process where a hand vein is catheterized to collect blood samples and intravenous lines are used to infuse glucose, saline, insulin, phenylalanine and amino acid solutions at at pre-specified times/rates. The mean GIR was calculated as the rate per kilograms of fat-free mass (FFM) during 4 hours of steady-state (hours 4-8 of the 8 hour clamp) reported as micromols/kilogram of FFM per minute. The FFM was measured by dual-energy x-ray absorptiometry (DEXA) scan. Insulin was infused with 5% essential amino acid solution (3mL/kg of FFM/hour) to prevent the insulin-dependent decrease of amino acids during insulin infusion.
Time Frame: Baseline, 3 months
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: micromols/kg of FFM/minute
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
micromols/kg of FFM/minute | 17.95 (8.60) | 1.68 (7.56)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in Fasting Blood Glucose Level
Description: Glucose (sugar) was measured in the blood and reported in milligrams per deciliter (mg/dL).
Time Frame: Baseline, 3 months
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
mg/dL | -19.96 (14.02) | 8.39 (22.51)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: HbA1c is a measure of average blood sugar levels over the preceding 3 month period. HbA1c was measured by ion-exchange chromatography and reported as a percentage.
Time Frame: Baseline, 3 months
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
percentage | -0.35 (0.40) | 0.19 (0.60)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change From Baseline in Insulin Levels
Description: Insulin levels in the blood were measured by immunoenzymatic assay and reported in micro International Units per milliliter (mcIU/mL).
Time Frame: Baseline, 3 months
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: microIU/mL
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
microIU/mL | -8.13 (7.47) | 1.38 (3.29)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline in Lipid Profile
Description: Change in lipids were measured by the change from baseline to 3 months of triglycerides, high-density lipoprotein cholesterol (HDL-C) and non-high-density lipoprotein cholesterol (non-HDL-C). All were reported in milligrams/deciliter (mg/dL).
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
mg/dL
  Triglycerides | -15.58 (32.67) | 17.77 (28.86)
  HDL-C-Cholesterol | 4.33 (6.75) | -0.31 (3.90)
  Non-HDL-Cholesterol | -7.50 (15.29) | 4.62 (17.76)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; P-value is for comparison between groups of the mean change in triglyceride levels; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Insulin Sensitizer Therapy vs Placebo; P-value is for comparison between groups of the mean change in HDL-C levels; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Insulin Sensitizer Therapy vs Placebo; P-value is for comparison between groups of mean change in non-HDL-C levels; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change From Baseline in the Thrombotic Biomarker Fibrinogen
Description: Fibrinogen was measured by thrombin clotting rate assay (Beckman Coulter, Inc. Brea, California) and reported in milligrams/deciliter (mg/dL).
Time Frame: Baseline, 3 months
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
mg/dL | 14.00 (71.24) | -18.62 (62.91)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change From Baseline in the Thrombotic Biomarker Plasminogen Activator Inhibitor-1 (PAI-1)
Description: PAI-1 was measured by enzyme-linked immunosorbent assay (Diagnostica Stago Inc., Parsippany, New Jersey) and reported in nanograms per milliliter (ng/mL).
Time Frame: Baseline, 3 months
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
ng/mL | -34.17 (25.35) | 8.15 (30.78)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change From Baseline in the Inflammatory Biomarker Interleukin 6 (IL-6)
Description: IL-6 is an inflammatory cytokine and reported in picograms per deciliter (pg/dL).
Time Frame: Baseline, 3 months
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
pg/mL | -0.99 (1.44) | -1.42 (4.84)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change From Baseline in the Inflammatory Biomarker C-Reactive Protein (CRP)
Description: CRP is an inflammatory cytokine and is reported in milligrams per deciliter (mg/dL).
Time Frame: Baseline, 3 months
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
mg/dL | -0.19 (0.22) | -0.15 (0.53)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change From Baseline in Inflammatory Biomarker Tumor Necrosis Factor-alpha (TNF-α)
Description: TNF-α is an inflammatory cytokine and is reported in picograms/milliliter (pg/mL).
Time Frame: Baseline, 3 month
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
pg/mL | -0.13 (0.21) | 0.18 (0.37)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change From Baseline in the Inflammatory Biomarker Adiponectin
Description: Adiponectin is an anti-inflammatory cytokine and is reported in milligrams per milliliter (mg/mL).
Time Frame: Baseline, 3 months
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
mg/mL | 9.10 (5.22) | 0.46 (0.92)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

12. Other Pre Specified Outcome: Change From Baseline in Body Mass Index
Description: Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The body mass index is an indication if a person is at a suitable weight for his height on an approximation of body fat.
Time Frame: Baseline, 3 months
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
kg/m^2 | 0.37 (0.62) | -0.21 (0.40)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney)

13. Other Pre Specified Outcome: Change From Baseline in Body Fat
Description: Body fat is reported as a percentage of body weight.
Time Frame: Baseline, 3 months
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
percentage of body weight | 1.73 (3.08) | -0.01 (1.44)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)

14. Other Pre Specified Outcome: Change From Baseline in Fat-Free Mass (FFM)
Description: FFM was measured using dual energy x-ray absorptiometry (DEXA) scans and is reported in kilograms (kg).
Time Frame: Baseline, 3 months
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Insulin Sensitizer Therapy | Placebo
Number analyzed (Participants) | 12 | 13
kilograms | -1.13 (2.81) | -0.34 (1.28)
Statistical Analysis 1: Comparison: Insulin Sensitizer Therapy vs Placebo; Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Insulin Sensitizer Therapy | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No